CLINICAL TRIAL: NCT05128396
Title: Successful Aging and Enrichment (SAGE): Effects of Environmental Stimulation on Cognitive Health and Neuroplasticity
Brief Title: Successful Aging and Enrichment (SAGE)
Acronym: SAGE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Linnaeus University (Other)
Responsible Party: Principal Investigator, Kirk Daffner, MD, Chief, Division of Cognitive and Behavioral Neurology, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 2013P002266
Record Dates: First submitted 2021-10-28; First posted 2021-11-22 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Cognitive Health; Healthy Aging
Keywords: aging; physical activity; cognitive stimulation; neural plasticity; mindfulness
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cognitive Training using Cogmed (Active Comparator): Subjects will complete computerized cognitive training with varying degrees of difficulty over 5 weeks.
  Interventions: Behavioral: Cognitive Stimulation
- Awareness (mindfulness) training (Active Comparator): Subject participate in mindfulness training. The meditation and tasks will become increasingly more self-directed over the 5 weeks; the degree of guidance will decrease to keep the subjective effort approximately constant and moderately challenging through the 5 weeks.
  Interventions: Behavioral: Mindfulness training
- Physical Exercise Training Using an Interactive Video Platform (Active Comparator): Subjects will participate in a structured physical exercise training program that aims to progressively increase their level of activity over the 5 week training period.
  Interventions: Behavioral: Physical Activity
- Low Level of Cognitive Training Using the Cogmed Program (Placebo Comparator): Subjects will complete the same computerized training as the active cognitive arm over the course of 5 weeks, but the main difference is that for the control group task difficulty will remain at the same low starting level, rather than increasing over time.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Cognitive Stimulation — During the initial session, a member of the research team will visit the subject's home and introduce the subject to the Cogmed training program (www.cogmed.com). Individuals will start at the same low difficulty level. As training proceeds, task difficulty will be individually adjusted based on performance by increasing/decreasing the number of items individuals have to remember, such that a participant reaches approximately 60% correct per day for each task. Each training session will start at the task difficulty level where the participant ended in the previous session. Performance and reaction time data will be continuously recorded while subjects are doing the task, and these data will be sent via the internet to the research team after each session. A member of the research team will communicate with each subject on a weekly basis (via phone call or email) to provide feedback and address any questions or concerns.
  Arms: Cognitive Training using Cogmed
Behavioral: Mindfulness training — The mindfulness meditations will be narrated by one guide and the tasks will be narrated by a different guide. We will have 7 mindfulness tasks in total, whose order of presentation will be counterbalanced across sessions: 1. mindful observing of place, 2. mindful eating, 3. mindful observing of object, 4. mindful observing of person, 5. mindful walking, 6. mindful listening, and 7. mindful writing with the non-dominant and dominant hand.
  At the end of each session, participants will write brief reflections stored via the website (e.g., an estimate of the amount of time subjects experienced their thoughts as wandering) both as an integral part of the mindfulness process and as a means of increasing the likelihood that subjects fully participate in each session. Each session will be structured as follows: Login, Mindfulness Meditation Session, Mindfulness Task 1, Mindfulness Task 2, Mindfulness Task 3, Write Log Reflection, Logout.
  Arms: Awareness (mindfulness) training
Behavioral: Physical Activity — Aerobic exercises will include relatively low impact activities like walking, jogging, or running in place, which will aim to put limited demands on balance. Each exercise will be explained and demonstrated in the video. All exercises can be done standing, sitting, or next to a chair that provides balance support as demonstrated in the videos. After the first session, for each subsequent session the difficulty level will start at one level below the previous session's average difficulty level (e.g. if they exercise at the most difficult level for most of the time during one session, the next session will start at the medium difficulty level). Each exercise will be explained and demonstrated in the video.
  Arms: Physical Exercise Training Using an Interactive Video Platform
Behavioral: Control Group — Individuals in the control group will participate in the same computerized Cogmed training program as described above. The main difference is that for the control group task difficulty will remain at the same low starting level, rather than increasing over time. The instructions given to subjects will be identical to the ones used in the cognitive training intervention.
  Arms: Low Level of Cognitive Training Using the Cogmed Program

SUMMARY:
Progress has been made in understanding the impact of different kinds of structured intervention programs in improving cognitive processing and performance in older adults, and in determining whether there is electrophysiological evidence for neuroplasticity in individuals over the age of 65.

DETAILED DESCRIPTION:
Study Procedures

Pre-Intervention Assessment The initial screening evaluation will take place over two half-day sessions, each lasting 3 to 3.5 hours in a designated room in the Laboratory of Healthy Cognitive Aging, Center for Brain/Mind Medicine, Brigham and Women's Hospital (BWH), 221 Longwood Avenue, Boston, Massachusetts (MA).

The sessions can be completed over one or two days, depending on the subject's preference.

Pre-Intervention Assessment Session 1 The first session will include completion of informed consent, a medical history, demographic information, including socioeconomic status (SES), survey questionnaires, and tests of visual acuity.

Screening Evaluation (for inclusion/exclusion)

Cognitive Screen

* The Mini-Mental State Examination (MMSE), a broad cognitive test on memory, spatial ability, memory and orientation, commonly used to screen for cognitive impairment
* American National Adult Reading Test (AmNART), a test of word pronunciation that provides an estimated IQ
* Logical Memory I and II, Wechsler Memory Scale-Third Edition, a test of verbal memory
* Boston Naming Test (Short-form, 15-items), a test of confrontation naming.

Depression Screen Geriatric Depression Scale

Neurological/Physical Evaluation Subjects will undergo a structured neurological examination. Height and weight will be obtained to calculate BMI. Visual acuity will be measured (Snellen wall chart).

Gait

Gait will be assessed through a procedure in which subjects walk 10 meters under two conditions:

1. Single task (walking at a comfortable pace)
2. Dual task (walking at a comfortable pace while simultaneously counting backwards by 3's, beginning with a 3 digit number told to the subject)

Every trial involving serial 3's will start from a different three digit number to reduce learning effects.

Subjects will be given an opportunity to carry out an untimed practice trial. Under the dual task condition, subjects will be instructed to perform as well as possible on both tasks (i.e., no specified prioritization). Each condition will be done 2 times, with the order counterbalanced across subjects. The first and last meter (gait start up and slow down) will not be counted in the measurements.

Time to walk 8 meters and number of steps taken will be measured. Under the dual task, investigators will also track how many numbers are generated while carrying out the serial 3's task (both correct and incorrect responses). In addition, the single task of counting backwards by 3's for 20 seconds will be tested twice in a seated position (once prior to and once after the gait testing).

Informant Questionnaire Subjects will select someone who knows them well (family member or friend) to complete a set of questionnaires. One questionnaire will provide information about a person's level of functioning (based on the Clinical Dementia Rating Scale), and another will inquire about a person's level of engagement (Apathy Scale). e questionnaires will be enclosed with a letter explaining how to complete the forms. The investigators will provide a stamped, addressed envelope to return the questionnaires to us. A backup plan will be to mail these materials directly to the informant selected. This would occur if the materials were misplaced or if the subject requests us to do so.

ELIGIBILITY:
Inclusion Criteria:

1. Be 65 or older
2. Have ≥ 8 years of education
3. Be sufficiently fluent in the English language to understand instructions and perform the neuropsychological tests (as the purpose of the project is to study healthy aging)
4. Score above levels indicating possible cognitive impairment on the Mini Mental State Exam (MMSE) (≥ 26)
5. Have an estimated intelligence quotient (IQ) score ≥ 90 based on the American National Reading Test (AmNART)
6. Have a score within 2 standard deviations (SD) of the age-appropriate mean on the short form of the Boston Naming Test
7. Have a score within 2 SD of the age-appropriate mean on the Logical Memory Subtest of the Wechsler Memory Scale-Third Edition

Exclusion Criteria:

1. History of Central Nervous System (CNS) diseases or major psychiatric disorders based on Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria
2. Score of greater than 10 on the Geriatric Depression Scale
3. Corrected visual acuity worse than 20-50 as tested by a Snellen wall chart
4. Severe hearing disability that would interfere with their ability to participate in the experiments (e.g., to hear instructions and participate in cognitive testing)
5. Medical conditions (e.g., heart or pulmonary disease) that would prevent them from participating in the physical exercise training program
6. Evidence of substantial functional decline based on interview questions and completion of a questionnaire based on the Clinical Dementia Rating Scale by an informant who knows the subject well

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cambridge Neuropsychological Test Automated Battery (CANTAB), a computerized assessment of cognitive functions | Baseline
  * CANTAB Paired Associate Learning (PAL) - assesses visual memory and new learning
  * CANTAB Attention Switching Task (AST) - measures cued attentional set-shifting
  * CANTAB Reaction Time (RTI) - measures speed of response to visual target when the stimulus is either predictable (simple RT) or unpredictable (choice RT)
  * CANTAB Spatial Span (SSP) - assesses working memory
  * CANTAB One Touch Stockings of Cambridge (OTS) - a test of non-verbal reasoning
Cambridge Neuropsychological Test Automated Battery (CANTAB), a computerized assessment of cognitive functions | End of Study - 5 weeks post-baseline
  * CANTAB Paired Associate Learning (PAL) - assesses visual memory and new learning
  * CANTAB Attention Switching Task (AST) - measures cued attentional set-shifting
  * CANTAB Reaction Time (RTI) - measures speed of response to visual target when the stimulus is either predictable (simple RT) or unpredictable (choice RT)
  * CANTAB Spatial Span (SSP) - assesses working memory
  * CANTAB One Touch Stockings of Cambridge (OTS) - a test of non-verbal reasoning
Trail Making Test A | Baseline
  Tests of visual attention and task switching Timed task - Max time allotted: 150 seconds
Trail Making Test A | End of Study - 5 weeks post-baseline
  Tests of visual attention and task switching Timed task - Max time allotted: 150 seconds
Trail Making Test B | Baseline
  Tests of visual attention and task switching Timed task - Max time allotted: 300 seconds
Trail Making Test B | End of Study - 5 weeks post-baseline
  Tests of visual attention and task switching Timed - Max time allotted: 300 seconds
Digit Symbol Coding, Weschler Adult Intelligence Scale (WAIS-IV) | Baseline
  A test of processing speed 90 seconds allowed - Higher scores indicate faster processing speed Maximum Score: 91 Minimum Score: 0
Digit Symbol Coding, Weschler Adult Intelligence Scale (WAIS-IV) | End of Study - 5 weeks post-baseline
  A test of processing speed 90 seconds allowed - Higher scores indicate faster processing speed Maximum Score: 91 Minimum Score: 0
Controlled Oral Word Association Test (COWAT) | Baseline
  A test of verbal retrieval and word generation Total score is measured by calculating the total number of acceptable words produced for all three letters.
Controlled Oral Word Association Test (COWAT) | End of Study - 5 weeks post-baseline
  A test of verbal retrieval and word generation Total score is measured by calculating the total number of acceptable words produced for all three letters
Categorical Fluency | Baseline
  A test of rapid retrieval of semantic knowledge Scored by counting the number of correct unique semantic category items produced
Categorical Fluency | End of study - 5 weeks post-baseline
  A test of rapid retrieval of semantic knowledge Scored by counting the number of correct unique semantic category items produced

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Feng NC, Ryan E, Kidane M, Tusch ES, McFeeley BM, Carlsson R, Mohammed AH, Hakansson K, Daffner KR. Feasibility of an at-home, web-based, interactive exercise program for older adults. Alzheimers Dement (N Y). 2019 Nov 22;5:825-833. doi: 10.1016/j.trci.2019.10.005. eCollection 2019. PMID 31799367
- [Background] Ledreux A, Hakansson K, Carlsson R, Kidane M, Columbo L, Terjestam Y, Ryan E, Tusch E, Winblad B, Daffner K, Granholm AC, Mohammed AKH. Differential Effects of Physical Exercise, Cognitive Training, and Mindfulness Practice on Serum BDNF Levels in Healthy Older Adults: A Randomized Controlled Intervention Study. J Alzheimers Dis. 2019;71(4):1245-1261. doi: 10.3233/JAD-190756. PMID 31498125
- [Background] Simon SS, Tusch ES, Feng NC, Hakansson K, Mohammed AH, Daffner KR. Is Computerized Working Memory Training Effective in Healthy Older Adults? Evidence from a Multi-Site, Randomized Controlled Trial. J Alzheimers Dis. 2018;65(3):931-949. doi: 10.3233/JAD-180455. PMID 30103334
- [Background] Tusch ES, Alperin BR, Ryan E, Holcomb PJ, Mohammed AH, Daffner KR. Changes in Neural Activity Underlying Working Memory after Computerized Cognitive Training in Older Adults. Front Aging Neurosci. 2016 Nov 8;8:255. doi: 10.3389/fnagi.2016.00255. eCollection 2016. PMID 27877122
- [Background] Hakansson K, Ledreux A, Daffner K, Terjestam Y, Bergman P, Carlsson R, Kivipelto M, Winblad B, Granholm AC, Mohammed AK. BDNF Responses in Healthy Older Persons to 35 Minutes of Physical Exercise, Cognitive Training, and Mindfulness: Associations with Working Memory Function. J Alzheimers Dis. 2017;55(2):645-657. doi: 10.3233/JAD-160593. PMID 27716670
- [Background] Simon SS, Tusch ES, Holcomb PJ, Daffner KR. Increasing Working Memory Load Reduces Processing of Cross-Modal Task-Irrelevant Stimuli Even after Controlling for Task Difficulty and Executive Capacity. Front Hum Neurosci. 2016 Aug 3;10:380. doi: 10.3389/fnhum.2016.00380. eCollection 2016. PMID 27536226

DOCUMENTS (1):
  • Study Protocol (2014-06-04): https://cdn.clinicaltrials.gov/large-docs/96/NCT05128396/Prot_000.pdf